CLINICAL TRIAL: NCT06564129
Title: Characteristics and Prehospital Triage of Anterior Large Vessel Occlusion Stroke Based on EEG
Brief Title: Prediction of Anterior Circulation Large Vessel Occlusion Stroke With EEG
Status: Not yet recruiting | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Junwei Hao, MD, Characteristics and prehospital triage of anterior large vessel occlusion stroke based on EEG, Xuanwu Hospital, Beijing
Other Study IDs: XMEC-2024-01
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Anterior Large Vessel Occlusion Stroke
Keywords: anterior large vessel occlusion stroke; electroencephalography; prehospital triage
MeSH Terms: interventions — Electroencephalography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: electroencephalography — Fifty-nine EEG electrodes conforming to international standard points were placed using a saline electrode EEG cap (Gelfree, Prysmian, China), and an accompanying portable multimodal EEG acquisition system (Neurohub, Prysmian, China) was used. EEG data were collected using collect software (Brycon, China).

SUMMARY:
This study is designed to evaluate the accuracy of saline electrode EEG in the prehospital diagnosis of LVO-a stroke.

DETAILED DESCRIPTION:
This is a multicenter, prospective, observational study,which will screen a total of 1194 patients in the participating centers during the period of June 1, 2024-December 31, 2025, and record single scalp EEG signals with eyes open at rest in the lying position of the patients using a non-invasive EEG acquisition device, and collect clinical data.

ELIGIBILITY:
Inclusion Criteria:

* Phase I.1.Acute ischemic stroke caused by occlusion of the anterior circulation (intracranial origin of the internal carotid artery or proximal middle cerebral artery (M1/M2)) confirmed by CTA, MRA or DSA (diagnosis in accordance with the "Chinese Guidelines for the Diagnosis and Treatment of Acute Ischemic Stroke 2023")；2. Patient age ≥18 years；3: Last normal time to EEG acquisition time ≤ 72 hours；4: Signed informed consent.

Phase II-III

1. Diagnosed by a healthcare professional as a suspected acute stroke patient or a known acute stroke patient
2. Patient age ≥18 years
3. Last normal time to EEG acquisition time ≤ 24 hours
4. Signed informed consent

Exclusion Criteria:

1. Wounds in the area of electrode cap placement or active infection in the scalp;
2. Patients who do not cooperate with the EEG examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients with suspected stroke or known stroke were included in the study
Sampling Method: Non-Probability Sample
Enrollment: 1194 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Saline electrode EEG characteristics: area under the ROC curve for theta/alpha ratio; | 24 hours
  Accuracy of theta/alpha ratio of electroencephalographic features for the diagnosis of large vessel occlusion
  Accuracy of theta/alpha ratio of electroencephalographic features for the diagnosis of anterior large vessel occlusion stroke

SECONDARY OUTCOMES:
Other EEG features including relative δ, θ, α power, δ/α ratio, δ+θ/α+β ratio, pdBSI, and WPLI diagnostic accuracy for LVO-a; | 24 hours
  ROC curves were plotted for each EEG data feature predicting LVO-a, and sensitivity, specificity, PPV, and NPV were calculated at the optimal cutoff value.
Logic and technical feasibility of saline electrode EEG in ambulance for suspected stroke patients by paramedics; | 24 hours
  Remove EEG data artifacts and report the percentage of EEG data available for analysis for each patient
Development of one or more new algorithms for optimal diagnosis of LVO-a based on EEG data | 24 hours
  ROC curves for predicted LVO-a based on this algorithm were plotted and sensitivity, specificity, PPV and NPV were calculated at the optimal cutoff value.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Beijing, Beijing, Beijing Municipality, China